CLINICAL TRIAL: NCT02390076
Title: Influence of Low-Level Light Therapy on Attention Bias Modification and Mood Change in Dysphoric Individuals
Brief Title: Behavioral Study of Effects of Low-Level Light Therapy on Mood and Reaction Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seth Disner (Other)
Responsible Party: Sponsor-Investigator, Seth Disner, Doctoral Candidate, University of Texas at Austin
Organization: University of Texas at Austin (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMHR-0001
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Left active LLLT (Active Comparator): Active LLLT targeting the left forehead Attention Bias Modification Left low level light therapy
  Interventions: Device: Left Low Level Light Therapy; Other: Attention bias modification
- Right active LLLT (Active Comparator): Active LLLT targeting the right forehead Attention Bias Modification Right low level light therapy
  Interventions: Other: Attention bias modification; Device: Right Low Level Light Therapy
- Sham LLLT (Sham Comparator): Sham LLLT targeting the right forehead Attention Bias Modification Sham low level light therapy
  Interventions: Other: Attention bias modification; Device: Sham Low Level Light Therapy

INTERVENTIONS:
Device: Left Low Level Light Therapy — Administration of left LLLT consists of applying light of a specific wavelength (1064 nanometers) using a laser diode, the CG-5000 high density laser (Cell Gen Therapeutics, LLC). Left LLLT will target the left forehead. The diameter parameters of stimulation are the same that showed psychologically beneficial effects in Schiffer et al. (2009). At the power level described, the energy emitted by the CG-5000 at this setting is one quarter of the skin MPE (0.250 W/cm2), exposure to it is not deemed harmful to tissue, and it causes no detectable physical damage and negligible heat.
  Other Names: Transcranial laser stimulation
  Arms: Left active LLLT
Other: Attention bias modification — The task will consist of a modified dot-probe paradigm. A pair of stimuli depicting a negative word and a neutral word will be presented, randomly located to the right and left side of the computer screen. The words will be presented for 1000 ms. The words will then disappear and a dot-probe will appear in the center of the screen location of one of the words (i.e., O or Q). This probe will appear on the screen until the participant presses one of two response buttons to indicate the identity of the probe. The presentation of the probe will be staggered to maximize attention for the neutral stimulus. Latency and accuracy of the button press responses are recorded by the computer.
  Other Names: Cognitive bias modification
Device: Right Low Level Light Therapy — Administration of right LLLT consists of applying light of a specific wavelength (1064 nanometers) using a laser diode, the CG-5000 high density laser (Cell Gen Therapeutics, LLC). Right LLLT will target the right forehead. The diameter parameters of stimulation are the same that showed psychologically beneficial effects in Schiffer et al. (2009). At the power level described, the energy emitted by the CG-5000 at this setting is one quarter of the skin MPE (0.250 W/cm2), exposure to it is not deemed harmful to tissue, and it causes no detectable physical damage and negligible heat.
  Other Names: Transcranial laser stimulation
  Arms: Right active LLLT
Device: Sham Low Level Light Therapy — Administration of sham LLLT is designed to resemble active LLLT from the participant's perspective, but uses a dosage markedly below the minimal necessary threshold to elicit a response.
  Other Names: Transcranial laser stimulation
  Arms: Sham LLLT

SUMMARY:
The goal of this project is to use low-level light therapy (LLLT) to enhance neural metabolism in the prefrontal cortex of humans, and measure the effects of LLLT on attentional bias change following a single session of attention bias modification (ABM). LLLT is non-invasive, therapeutically beneficial, and promotes a wide range of biological effects including enhancement of energy production, gene expression and prevention of cell death. Previous research has indicated that human participants show a beneficial psychological effect, including improved mood and greater sustained attention, following a single treatment of LLLT to the forehead. ABM is a computer-based cognitive task designed to decrease the mood-congruent negative attentional bias frequently observed in depressed and dysphoric individuals. Previous ABM studies have led to decrease in clinical symptoms relative to a control condition. This study will explore whether the effects of LLLT on mood and attention could improve the potency of ABM, leading to greater attention change and greater improvement of mood relative to sham LLLT.

DETAILED DESCRIPTION:
Low-level light therapy constitutes a novel intervention shown to regulate neuronal function in cell cultures, animal models, and clinical conditions. The Gonzalez-Lima lab has previously shown that low-level light therapy can increase mitochondrial cytochrome oxidase activity, which can provide neuroprotection against toxicity and can improve the aerobic capacity of other tissue such as skeletal muscle. This suggests that the oxidative metabolism of tissue exposed to LLLT is enhanced. LLLT treatments also appear to have in vivo transcranial neurochemical effects that involve metabolic-enhancing and antioxidant systems; it is a non-invasive technique that has been used in humans to stimulate the brain as an antidepressant treatment, to alleviate muscle fatigue and enhance recovery, and to increase sustained attention during cognitive tasks. These LLLT treatments have thus been proven to be not just safe but actually beneficial in humans. Collectively, these data imply that LLLT could be used as an inexpensive, noninvasive approach to boost blood flow and energy consumption in the brain and other tissues, as well as provide neuroprotection against neurological conditions which may be related to mitochondrial dysfunction. This research could ultimately lead to the development of non-invasive, non-pharmacologic, therapeutic, cytoprotective and performance-enhancing interventions in both healthy humans and in those in need of rehabilitation efforts under conditions where neuromuscular function and movement are compromised, as well as treating neurobiological disorders in which metabolic dysfunction plays an underlying causal role, such as depression and post-traumatic stress disorder.

The therapeutic use of red to near-infrared light wavelengths is based on the principle that certain molecules in living systems absorb photons and trigger signaling pathways in response to light. In biologic tissues, absorption and scattering of light (which would render it ineffective as a treatment) are maximal at wavelengths below 600 nanometers, and water absorbs light at wavelengths greater than 1150 nanometers. Thus, there is a "wavelength window" for biologic stimulation that covers the red to near-infrared light spectrum (between 600 and 1150 nm).

Early results suggest that LLLT may have significant promise in the treatment of clinical disorders. Prior work found that a single LLLT treatment to the forehead resulted in an increased cerebral blood flow and significant beneficial effect in patients with major depression and anxiety. Previous research conducted in the Gonzalez-Lima lab showed that healthy human subjects receiving LLLT showed significantly higher positive affect at two week follow-up sessions relative to subjects in the "placebo-light" condition. Importantly, no adverse side effects were found in subjects for either study, either immediately after the initial treatment, or at two or four weeks post-treatment. The investigators plan to follow the LLLT treatment protocol from these two studies, immediately prior to running subjects through the ABM procedure.

ABM is a technique designed to modify attentional bias, a cognitive factor that has been theorized to underlie the onset and maintenance of Major Depressive Disorder. ABM is built on the framework of the standard dot-probe task, wherein two valenced stimuli are presented side-by-side, and then followed by a target probe behind one of the stimuli. The difference in response time between probes directly behind a stimuli relative to probes on the opposite side of the stimuli can be used to operationalize attentional bias for that particular valence of stimuli. ABM uses a conditioning approach to shift this bias by staggering the frequency of probe distribution in favor of one specific valence. Eventually, participants are expected to preferentially process the favored valence of stimuli, leading to a shifting of attentional bias.

This placebo-controlled study will measure whether LLLT influences the efficacy of ABM on measures of biased attention and dysphoria. Participants will be randomized to receive either active or placebo LLLT, and will then undergo an ABM procedure designed to decrease attention towards negative environmental stimuli (measured using a variant of the dot-probe task). The combination of LLLT and ABM will take place over two sessions (two days apart), and will be followed by one and two week follow-up periods to assess mood change. The investigators hypothesize that participants who receive the active LLLT will show greater change in attentional bias following ABM and greater decrease in dysphoric symptoms during follow-up compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old,
* English as first language,
* baseline CES-D score > 16.

Exclusion Criteria:

* active neurological condition (such as epilepsy or stroke).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Left Active LLLT: Active LLLT targeting the left forehead Attention Bias Modification Left low level light therapy
  Left Low Level Light Therapy: Administration of left LLLT consists of applying light of a specific wavelength (1064 nanometers) using a laser diode, the CG-5000 high density laser (Cell Gen Therapeutics, LLC). Left LLLT will target the left forehead.
  Attention bias modification: The task will consist of a modified dot-probe paradigm. A pair of stimuli depicting a negative word and a neutral word will be presented, randomly located to the right and left side of the computer screen. The words will be presented for 1000 ms. The words will then disappear and a dot-probe will appear in the center of the screen location of one of the words (i.e., O or Q). This probe will appear on the screen until the participant presses one of two response buttons to indicate the identity of the probe. Latency and accuracy of the button press responses are recorded by the computer.
- Right Active LLLT: Active LLLT targeting the left forehead Attention Bias Modification Right low level light therapy
  Right Low Level Light Therapy: Administration of left LLLT consists of applying light of a specific wavelength (1064 nanometers) using a laser diode, the CG-5000 high density laser (Cell Gen Therapeutics, LLC). Left LLLT will target the right forehead.
  Attention bias modification: The task will consist of a modified dot-probe paradigm. A pair of stimuli depicting a negative word and a neutral word will be presented, randomly located to the right and left side of the computer screen. The words will be presented for 1000 ms. The words will then disappear and a dot-probe will appear in the center of the screen location of one of the words (i.e., O or Q). This probe will appear on the screen until the participant presses one of two response buttons to indicate the identity of the probe. Latency and accuracy of the button press responses are recorded by the computer.
- Sham LLLT: Sham LLLT targeting the right forehead Attention Bias Modification Sham low level light therapy
  Attention bias modification: The task will consist of a modified dot-probe paradigm. A pair of stimuli depicting a negative word and a neutral word will be presented, randomly located to the right and left side of the computer screen. The words will be presented for 1000 ms. The words will then disappear and a dot-probe will appear in the center of the screen location of one of the words (i.e., O or Q). This probe will appear on the screen until the participant presses one of two response buttons to indicate the identity of the probe. Latency and accuracy of the button press responses are recorded by the computer.
  Sham Low Level Light Therapy: Administration of sham LLLT is designed to resemble active LLLT from the participant's perspective, but uses a dosage markedly below the minimal necessary to elicit a physiological response.
Period: Overall Study
Arm/Group | Left Active LLLT | Right Active LLLT | Sham LLLT
Started | 18 | 18 | 15
Completed | 16 | 17 | 11
Not Completed | 2 | 1 | 4
Not completed — Lost to Follow-up | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Left Active LLLT | Right Active LLLT | Sham LLLT | Total
Number analyzed (Participants) | 18 | 18 | 15 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.22 (1.48) | 18.72 (0.89) | 20.33 (5.29) | 19.37 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 10 | 31
  Male | 9 | 6 | 5 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 6 | 3 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 9 | 9 | 12 | 30
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 15 | 51

OUTCOME MEASURES:

1. Primary Outcome: Presence and Severity of Depressive Symptoms Assessed by Center for Epidemiologic Studies - Depression Scale (CES-D)
Description: The CES-D (Radloff, 1977) is a 20-item, self-report scale designed to assess the presence and severity of depressive symptoms over the past week. The total range is 0-80, with higher scores reflecting more severe depression symptoms. Outcome measure data table reflects clinical symptoms at 2 week follow-up.
Time Frame: At baseline, session 1, session 2, 1 week follow-up, and 2 week follow-up.
Measure: Mean (Standard Deviation); unit: units on a the CESD scale
Arm/Group | Left Active LLLT | Right Active LLLT | Sham LLLT
Number analyzed (Participants) | 18 | 18 | 15
units on a the CESD scale | 21.93 (10.15) | 22.5 (9.77) | 21.75 (8.45)

2. Secondary Outcome: Biased Attention for Emotional Stimuli Measured by the Dot Probe Task
Description: This task measures biased attention for emotional stimuli. In this task, two stimuli are presented at the same time. The investigators plan to present two words concurrently; one emotionally valenced word (positive or negative) and one neutral word. Two words appear on the screen for 1000 ms; the location of the emotional and neutral word varies randomly. Following the offset of the words, a subsequent target (i.e., O or Q) appears; the location of the target is randomized with the constraint that it must appear an equal number of times behind the emotional and neutral words. Each iteration of the dot probe task will include 96 trials, and will last approximately 7 minutes. Behavioral reaction times are recorded via a button push on the response box. Change in negative bias is calculated as mean bias value from the dot probe task at the end of session 2 minus the mean bias value calculated at the beginning of session 1.
Time Frame: Measure was administered at the beginning of session 1 and end of session 2.
Measure: Mean (Standard Deviation); unit: change in negative bias (ms)
Arm/Group | Left Active LLLT | Right Active LLLT | Sham LLLT
Number analyzed (Participants) | 18 | 18 | 15
change in negative bias (ms) | -24.15 (67.66) | 4.28 (31.43) | -3.08 (25.64)

ADVERSE EVENTS:
Time Frame: Participants were followed for two weeks after their initial enrollment.
Description: Participants were asked about any adverse events since their last study contact.
Arm/Group | Left Active LLLT | Right Active LLLT | Sham LLLT
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No